CLINICAL TRIAL: NCT00035893
Title: The Role of Ampligen in Strategic Therapeutic Intervention (STI) of Highly Active Anti-Retroviral Therapy (HAART): A Multi-Center, Randomized, Controlled Study of Ampligen Potentiation of the HAART-Free Interval.
Brief Title: The Role of Ampligen in Strategic Therapeutic Intervention (STI) of HAART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMP 720
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: HIV Seropositivity; HIV Infection
Keywords: treatment interruption; HIV Infections
MeSH Terms: conditions — HIV Seropositivity; HIV Infections | interventions — poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ampligen (Experimental): Ampligen (poly I-poly C12U) 200-400 mg IV infusions given twice weekly for 64 weeks.
  Interventions: Drug: poly I-poly C12U
- No Ampligen (No Intervention): No Ampligen administered for first 64 weeks

INTERVENTIONS:
Drug: poly I-poly C12U — 200-400 mg IV infusions 2x/week for 64 weeks
  Other Names: Ampligen; Rintatolimod
  Arms: Ampligen

SUMMARY:
This is an open-label, prospective, randomized, controlled study of the safety and efficacy including clinical, immunologic, and virologic assessments of adding Ampligen to a Strategic Therapeutic Intervention (STI) of HAART in patients with plasma HIV RNA < 50 copies/ml (PCR) and CD4 levels > 400.

ELIGIBILITY:
1. Adults at least 18 years of age.
2. CD4 cell count of > 400 cells.
3. Plasma HIV-1 RNA < 50 copies/ml on two occasions: one within the six weeks prior to starting Baseline and the other during Baseline.
4. History of virologic success with suppression of HIV RNA level < 50 copies/ml during the last nine months documented a minimum of two times during the last ten months or a minimum of three times during the last fifteen months while patient is receiving a HAART regiment. During the four months prior to starting Baseline, continuing through Baseline and the 64 week study period, the HAART regimen must remain unchanged and contain at least one of the following ten anti-retroviral drugs:

   * Abacavir (Ziagen)
   * Zidovudine (Retrovir) AZT
   * Zalcitabine (Hivid) ddC
   * Didanosine (Videx) ddl
   * Stavudine (Zerit) d4T
   * Efavirenz (Sustiva)
   * Indinavir (Crixivan)
   * Ritonavir (Norvir)
   * Nelfinavir (Viracept)
   * Amprenavir (Agenerase)

   Only one HIV plasma RNA level > 50, but < 100 copies/ml is permitted during the four month period immediately prior to starting Baseline.
5. Karnofsky performance status of at least 70.
6. The following laboratory parameters within 21 days prior to treatment:

   * Hemoglobin > 9.2 g/dL for men and > 8.9 g/dL for women;
   * Neutrophil count > 1000;
   * Platelet count > 75,000;
   * AST/ALT < 4.0 x upper limit of normal (ULN);
   * Serum creatinine < 1.5 x ULN or a creatinine clearance > 50 mL/min.
7. Ability and willingness to give written informed consent.
8. For females with child bearing potential: A negative serum pregnancy test within 14 days prior to randomization. Females of child bearing potential agree to use an effective means of contraception.
9. The patient must have completed any elective routine immunizations (including influenza vaccination) eight or more weeks prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
HAART-free time interval | HAART adherence questionnaire completed weekly
  To evaluate the potential effectiveness of Ampligen to increase the HAART-free time interval before HIV rebound during the STI of HAART.

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (10):
- United States (10):
  - Orange County Center for Special Immunology, Fountain Valley, California
  - AltaMed Health Services Corporation, Los Angeles, California
  - Circle Medical Center, Norwalk, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Julia Torres, MD, Fort Lauderdale, Florida
  - Allied Clinical Trials, Miami, Florida
  - Scott Ubillos, MD, Tampa, Florida
  - St. Michael's Medical Center, Newark, New Jersey
  - Christopher Lucasti, D.O., Somers Point, New Jersey
  - W. Chris Woodward, DO, Reading, Pennsylvania